CLINICAL TRIAL: NCT00548535
Title: Is Self-Reported Quality Assessment in Surgery Reliable?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Other Study IDs: DDI1007
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2007-10-24 (Estimated); Status verified 2007-10

CONDITIONS: Patients of Visceral- and Transplantation Surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Reliability of complication assessment

SUMMARY:
Aim of the study is to evaluate the reliability of self-reported surgical outcome by residents

* prospective assessment of postoperative complications done by residents using a validated five-scale complication classification
* simultanously, complications will be prospectively assessed in the same manner by an external clinical nurse
* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* All patients undergoing elective surgery

Exclusion criteria:

* Patients not undergoing surgery
* Patient in outpatient setting

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dindo, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland